CLINICAL TRIAL: NCT06742177
Title: Comparison of Bi-Level Erector Spinae Plane Block (ESPB) and Modified Thoraco Abdominal Plane Block (M-TAPA) in Laparoscopic Abdominal Surgery
Brief Title: Comparison of Bi-Level Erector Spinae Plane Block (ESPB) and Modified Thoraco Abdominal Plane Block (M-TAPA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Seyyid Furkan Kına, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0067
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Opioid Consumption; Numerical Rating Scale; Demographic Data
Keywords: Modified Thoraco Abdominal Block; Erector Spinae Plane Block; Abdominal surgery; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Bi-level ESPB (Active Comparator): The block procedure is performed immediately before surgery begins after general anesthesia induction, with the patient in the lateral decubitus position. For the block, sterile conditions are provided with USG, and the erector spinae muscle and vertebral process are visualized, and the in plane technique is used. The target vertebral level for bi-level ESPB is two levels, T5 and T7. The block needle is advanced in the caudo-cranial direction, and the potential area between the erector spinae muscle and the transverse process of the relevant vertebra is targeted. The block location is confirmed by injecting 2 ml of saline between the transverse process and the muscle. After the block location is confirmed, a total of 40 ml of 0.25% bupivacaine is applied, using 20 ml of 0.25% bupivacaine for a single level.
  Interventions: Procedure: Group Bi-level ESPB
- Group M-TAPA Block (Active Comparator): The procedure is performed in the supine position immediately before surgery after general anesthesia induction and the in plane technique is used. The transversus abdominis, internal oblique and external oblique muscles are identified at the costochondral angle in the sagittal plane under ultrasound guidance at the 10th costal margin. The block needle is advanced in the caudo-cranial direction and a deep angle is given with the probe in the sagittal direction to the costochondral angle at the edge of the 10th rib to visualize the lower surface of the costal cartilage in the midline. The block location is confirmed by injecting 2 ml of saline onto the transverse abdominis muscle under the 10th costal cartilage. After the block location is confirmed, 20 ml of 0.25% bupivacaine is used. This procedure is repeated for the opposite side and a total of 40 ml of 0.25% bupivacaine is used.
  Interventions: Procedure: Group M-TAPA block

INTERVENTIONS:
Procedure: Group Bi-level ESPB — The block procedure is performed immediately before surgery begins after general anesthesia induction, with the patient in the lateral decubitus position. For the block, sterile conditions are provided with USG, and the erector spinae muscle and vertebral process are visualized, and the in plane technique is used. The target vertebral level for bi-level ESPB is two levels, T5 and T7. The block needle is advanced in the caudo-cranial direction, and the potential area between the erector spinae muscle and the transverse process of the relevant vertebra is targeted. The block location is confirmed by injecting 2 ml of saline between the transverse process and the muscle. After the block location is confirmed, a total of 40 ml of 0.25% bupivacaine is applied, using 20 ml of 0.25% bupivacaine for a single level.
  Arms: Group Bi-level ESPB
Procedure: Group M-TAPA block — The procedure is performed in the supine position immediately before surgery after general anesthesia induction and the in plane technique is used. The transversus abdominis, internal oblique and external oblique muscles are identified at the costochondral angle in the sagittal plane under ultrasound guidance at the 10th costal margin. The block needle is advanced in the caudo-cranial direction and a deep angle is given with the probe in the sagittal direction to the costochondral angle at the edge of the 10th rib to visualize the lower surface of the costal cartilage in the midline. The block location is confirmed by injecting 2 ml of saline onto the transverse abdominis muscle under the 10th costal cartilage. After the block location is confirmed, 20 ml of 0.25% bupivacaine is used. This procedure is repeated for the opposite side and a total of 40 ml of 0.25% bupivacaine is used.
  Arms: Group M-TAPA Block

SUMMARY:
Laparoscopy is a surgical technique used for basic diagnosis and treatment. The advantages of laparoscopic techniques compared to open surgery have been demonstrated by studies. With the developing medicine and technology, minimally invasive approaches have been targeted in interventional procedures. In laparoscopic surgeries, access to the abdomen is provided with the help of a trocar and a temporary pneumoperitoneum is created with gas insufflation. Despite all these developments, even when laparoscopic techniques are used, postoperative pain is the most disturbing issue for patients. Postoperative pain can seriously reduce the quality of life in patients and acute pain can even trigger chronic pain syndromes. Epidural analgesia, paravertebral, erector spinae plane, intercostal nerve, transverse abdominis plane, external oblique, modified thoracoabdominal plane, rectus sheath block are used for anesthesia and analgesia during laparoscopic abdominal surgeries (LAS). In recent years, regional nerve blocks, including erector spinae plane block (ESPB) and modified thoraco-abdominal plane block (M-TAPA), have been applied for the treatment of pain in patients undergoing LAS due to various causes. ESPB was first described by Forero et al. in 2016 and has been frequently used for the treatment of acute pain in the postoperative period following abdominal surgeries. ESPB can be applied at any level from cervical to sacral, covering dermatomes appropriate for the surgical area under USG guidance. Cadaver studies for the ESPB mechanism have shown that local anesthetic spreads ipsilaterally and contralaterally and that it has analgesic efficacy both on the side where it is applied and on the opposite side. This peripheral nerve block, which is usually applied at a single level, can also be applied at bi-level. Studies have also shown that when ESPB is applied at bi-level, analgesic efficacy increases due to local anesthetic spread.

M-TAPA is a new peripheral nerve block technique defined by Tulgar et al. It has high analgesic efficacy in thoraco-abdominal surgery. It has been shown to be advantageous in upper umbilical surgeries by involving more dermatomes compared to the transverse abdominis plane block. Lateral and anterior branches of thoraco-abdominal nerves are blocked with M-TAPA. It provides analgesia in a wide area between T5 and T12 and can also be applied for LAS. In our clinic, Bi-level ESPB or M-TAPA is routinely applied to suitable patients after anesthesia induction, and intraoperative anesthesia is maintained with inhalation and intravenous anesthetic agents. Multimodal analgesia management has been adopted as postoperative analgesia management.

ELIGIBILITY:
Inclusion Criteria:

1-Patients over 18 years of age

2.Those with ASA score I-II-III

3.Those with body mass index (BMI) between 18-40

4.Patients who underwent LAS in the operating room with Bi-level ESPB or M-TAPA

Exclusion Criteria:

1. Those under 18 years of age
2. Those with ASA score IV and above
3. Those with advanced co-morbidities
4. Those with a history of bleeding diathesis
5. Patients with infection in the area where the block will be performed
6. Those with BMI below 18 and above 40
7. Patients who underwent surgery under emergency conditions

8- Patients with advanced liver and kidney failure

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative opioid consumption. | Intraoperative period
  Intraoperative opioid consumption will be recorded.

SECONDARY OUTCOMES:
Pain Scores | 24 hours after surgery
  Pain will be assessed using a numerical rating scale from 0 (no pain) to 10 (worst pain) at rest and during coughing. Pain assessment will be made at 1, 2, 6, 12, and 24 hours after surgery. The numerical rating scale is 10 (worst) severe, unbearable pain; 0 (best) no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Seyyid Furkan Seyyid Furkan, MD, Principal Investigator — Ankara Etlik City Hospital